CLINICAL TRIAL: NCT05383690
Title: Effects of Litebook EDGE™ Phototherapy on Academic Performance and Functional Brain Activity in Non-Depressed Adolescents
Brief Title: Effects of Litebook EDGE™ Phototherapy on Academic Performance and Brain Activity
Acronym: LiteBook
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: LiteBook Company Ltd (Unknown)
Responsible Party: Principal Investigator, Martin H Teicher, Research Psychiatrist, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016D003724
Record Dates: First submitted 2022-05-08; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Sleepiness, Daytime
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: Single arm, with independent variable being percent device use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bright Light Arm (Experimental): This is a one-arm study. Subjects will be provided with the LiteBook Edge™ (LiteBook Company LTD), which is a patented smart phone sized BLT device that provides 10,000 lux illumination at a recommended distance of 61 cm from an LED panel with peak spectral radiance in the blue color spectrum that closely corresponds to the peak spectral frequency (480 nm) of melanopsin photoreceptors that project to the suprachiasmatic nucleus and entrain the circadian clock (Hatori & Panda, 2010).
  Interventions: Device: LED bright light treatment device

INTERVENTIONS:
Device: LED bright light treatment device — Subjects will be instructed to use the bright light treatment device, as early as possible, for 30 minutes each morning. These devices will be equipped with monitoring electronics that will enable us to download their daily degree of use. Participants will also be provided with yellow-tinted blue light blocking glasses and will be instructed to wear them starting 2 hours before bedtime if they are viewing LED or liquid-crystal display screens.
  Other Names: LiteBook Edge™

SUMMARY:
As children pass through puberty the timing of their sleep-wake cycle shifts and they experience a strong urge to stay up and awaken late. High school typically starts early in the morning and a significant percentage of normal adolescents arrive at school each day with an insufficient amount of sleep, which can take a substantial toll on their academic performance. As the primary reason for insufficient sleep is a naturally occurring propensity to stay up later in the evening it seems plausible that bright light treatment (BLT) at the appropriate time may phase advance biological clocks and potentially reverse this problem. Hence, the investigators are testing the hypothesis that consistent morning use of a light emitting diode (LED) BLT device (LiteBook Edge™) by healthy adolescents will shift the phase of their sleep wake cycle and enable them to receive an increased amount of sleep during the school week and perform better on tests of attention and academic performance and evidence signs of improved alertness. Alternatively, BLT could potentially enhance alertness through other mechanisms, such as a direct arousing effect, without exerting a discernible effect on circadian phase or sleep duration.

DETAILED DESCRIPTION:
As children pass through puberty the timing of their sleep-wake cycle shifts and they experience a strong urge to stay up and awaken late. Hence, a large percentage of normal adolescents arrive at school each day with an insufficient amount of sleep, which can take a substantial toll on their academic performance.

A growing number of human studies show that sleep promotes learning and memory. Conversely, sleep deprivation has a negative impact on cognitive and behavioral functions. Relatively few studies have examined effects of sleep deprivation on cognitive performance in adolescents. In these studies, total sleep deprivation was associated with impaired memory performance and diminished computational speed, while, partial sleep deprivation was associated with deficits in reasoning and verbal creativity. For example, male adolescents sleeping more than 8 hours per day had significantly higher reasoning ability than their peers who slept for less than 8 hours per day. Some studies reported that simpler cognitive processes such as working memory and computational speed may not be significantly affected by a single night of sleep limited to 4 to 5 hours. However, even mild sleep restriction of an hour or more, when persistent across days, can lead to memory problems as severe as seen following total sleep deprivation.

The sensitivity of the adolescent brain to subtle sleep impairments was highlighted in a study where 12-14-year-olds were allowed to play stimulating computer games or watch television right before bedtime. This experience prolonged sleep latency, increased stage 2 sleep and reduced slow wave sleep. This modest degree of sleep restriction significantly impaired verbal memory consolidation Suboptimal sleep duration in adolescents was also associated with poor performance on a serial digit-learning test during morning testing sessions, but not in afternoon sessions. Between 58-68% of high school students surveyed in Ontario report that they feel "really sleepy" between 8 and 10 A.M. Thus, achievement in early morning classes may suffer the most in sleep-deprived adolescents.

Fortunately, sleep only needs to be extended by a modest amount to enhance cognition in children. Sadeh showed that performance on memory, attention and vigilance tasks in children improved significantly after 1 hour of sleep extension on three consecutive nights. Gais and Backhaus have also shown the beneficial effects of sleep on memory consolidation in children and adolescents.

Overall, there is compelling scientific evidence that schoolchildren, particularly adolescents, are chronically sleep deprived, that the degree of sleep restriction they experience exerts demonstrable effects on memory encoding, consolidation and processing speed, and that even a modest increase in sleep will result in measurable improvements in cognitive function. The primary reason that adolescents are sleep deprived is due to a naturally occurring phase delay in their biological clock, resulting in a propensity to stay up until late in the evening which is incompatible with the early rise times schools typically require. Light treatments at the appropriate time can phase advance the biological clock, potentially reversing this problem.

The hypothesis that the investigators propose to test is that consistent morning use of the Litebook Edge™ bright light therapy device, coupled with two-hour pre-bedtime use of blue-wave light blocking glasses while watching video screens will shift the circadian phase of the sleep-wake cycle of normal adolescents. This in turn will enable them to fall asleep earlier and to receive an increased amount of sleep during the school week. Consequently, they will awaken more readily, feel more awake during early classes, and will perform better on tests of academic performance, attention and working memory. Light therapy will enhance functional connectivity of prefrontal regions involved in attention. Degree of improvement in cognition, attention and functional and structural MRI measures will be directly related to average time spent each day activating (and presumably using) the device, which will be the independent variable in the statistical analyses.

This is a one-arm study, and all participants will receive active treatment. The device was designed to monitor degree of use and the primary statistical question is whether there is a significant association between degree of use and improvement in measures of wakefulness, alertness, and cognitive performance.

This approach of using duration of device activation as the independent variable, in a small preliminary study, provides several advantages over a two-arm studying comparing bright white light to either placebo red light or another type of mechanical device. First, effect size measures previously calculated assumed that subjects in both groups would use the device. There will likely be significant variability between subjects in degree of use and if only a fraction of subjects assigned the bright light device used it consistently then the overall impact would be weaker and possibly missed in a two-group analysis. Using duration of device operation will enable the investigators to compare subjects who used it to a considerable degree versus subjects who hardly use it at all and would likely provide a good estimate of how much benefit accrues from different degrees of use.

This is particularly important for the neuroimaging component. If the investigators compared active versus placebo devices, then only half of the neuroimaged subjects would receive the active device, which may leave the investigators comparing pre versus post effects in only 8-10 subjects. In this revised design all the neuroimaged sample (n = 16-20) would receive the active treatment making the pre-post comparisons stronger, especially when adjusted for duration of device activation.

Second, using duration of device activation as the independent variable will markedly facilitate recruitment. If the investigators used a placebo device, they would need to indicate in the informed consent that subjects may receive a placebo device, without revealing what the placebo is. Instead, the investigators can now indicate in the informed consent that all subjects will receive a device that they believe is biologically active and that no placebos will be used.

This also makes the protocol simpler as raters do not need to be kept blind to device type. All the investigators need to do is make sure that raters remain unaware of duration of device activation.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in school, drowsiness/sleepiness during morning classes which interferes to some degree with academic performance but able to wake up and be on time for said classes, willingness to use a device in the morning to enhance alertness, Intelligence Quotient greater than 80

Exclusion Criteria:

* Symptoms of psychiatric disorder on screening, current use of medications, home schooled, involved in morning activities, like athletics, that can alter morning alertness

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Beta electroencephalographic (EEG) activity | Baseline and week 4 (or last observation after baseline)
  Primary outcome measure one is the degree of increase in beta EEG activity, which is indicative of wakefulness and arousal. Change in beta EEG power will be compared to degree of use of the bright light treatment device.
Theta electroencephalographic (EEG) activity | Baseline and week 4 (or last observation after baseline)
  Primary outcome measure two is the degree of decease in theta EEG activity, which is indicative of drowsiness. Change in theta EEG power will be compared to degree of use of the bright light treatment device.
Sleep onset | Baseline and week 4 (or last observation after baseline)
  Primary outcome measure three is the change in actigraph-assessed sleep onset to an earlier hour. Change in sleep onset time will be compared to degree of use of the bright light treatment device.
Sleep duration | Baseline and week 4 (or last observation after baseline)
  Primary outcome measure four is the increase in actigraph-assessed sleep duration. Change in sleep duration will be compared to degree of use of the bright light treatment device.

SECONDARY OUTCOMES:
Errors of omission | Baseline and week 4 (or last observation after baseline)
  Errors of omission on the Quotient ADHD System provides a measure of inattention. These errors occur when a subject fails to respond to a target stimulus. Degree of reduction in errors of omission will be compared to degree of use of the bright light treatment device.
Response variability | Baseline and week 4 (or last observation after baseline)
  Variability in response speed on the Quotient ADHD System to target stimuli provides another measure of inattention. Degree of reduction in response variability will be compared to degree of use of the bright light treatment device.
Mathematical ability | Baseline and week 4 (or last observation after baseline)
  Participants will be tested on their ability to correctly solve as many complex math problems from high school placement exam as they can in 10 minutes. Degree of improvement will be compared to degree of use of the bright light treatment device.
Simple computational speed | Baseline and week 4 (or last observation after baseline)
  Fifty single digit addition and subtraction problems will be presented to participants using the Modified Walter Reed serial addition/subtraction task to assess computational speed. Degree of improvement will be compared to degree of use of the bright light treatment device.
Dentate gyrus volume | Baseline and week 4 (or last observation after baseline)
  The volume of the dentate gyrus, a portion of the hippocampal complex in the brain will be measured using magnetic resonance imaging. This brain region is involved in memory processes and can change in size in response to stress and sleep deprivation. Increase in dentate gyrus volume will be compared to degree of use of the bright light treatment device.
Sleep propensity | Baseline and week 4 (or last observation after baseline)
  Self-reported change in propensity to fall asleep in various situations will be assessed using the Epworth Sleepiness Scale. Degree of reduction in sleep propensity will be compared to degree of use of the bright light treatment.

OTHER OUTCOMES:
Functional connectivity during Go/No Go task | Baseline and week 4 (or last observation after baseline)
  Functional MRI imaging will be used to assess changes in the connectivity of prefrontal cortical regions during performance of a Go/No Go attention task to identify brain regions in which degree of increase in connectivity corresponds to degree of use of the bright light treatment device.

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Teicher, MD,PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backhaus J, Hoeckesfeld R, Born J, Hohagen F, Junghanns K. Immediate as well as delayed post learning sleep but not wakefulness enhances declarative memory consolidation in children. Neurobiol Learn Mem. 2008 Jan;89(1):76-80. doi: 10.1016/j.nlm.2007.08.010. Epub 2007 Oct 29. PMID 17911036
- [Background] Banks S, Dinges DF. Behavioral and physiological consequences of sleep restriction. J Clin Sleep Med. 2007 Aug 15;3(5):519-28. PMID 17803017
- [Background] Born J, Rasch B, Gais S. Sleep to remember. Neuroscientist. 2006 Oct;12(5):410-24. doi: 10.1177/1073858406292647. PMID 16957003
- [Background] Born J, Wagner U. Sleep, hormones, and memory. Obstet Gynecol Clin North Am. 2009 Dec;36(4):809-29, x. doi: 10.1016/j.ogc.2009.10.001. PMID 19944302
- [Background] Cajochen C. Alerting effects of light. Sleep Med Rev. 2007 Dec;11(6):453-64. doi: 10.1016/j.smrv.2007.07.009. Epub 2007 Nov 1. PMID 17936041
- [Background] Carskadon MA, Acebo C, Jenni OG. Regulation of adolescent sleep: implications for behavior. Ann N Y Acad Sci. 2004 Jun;1021:276-91. doi: 10.1196/annals.1308.032. PMID 15251897
- [Background] Carskadon MA, Harvey K, Dement WC. Sleep loss in young adolescents. Sleep. 1981 Sep;4(3):299-312. doi: 10.1093/sleep/4.3.299. PMID 7302461
- [Background] Carvalho-Mendes RP, Dunster GP, de la Iglesia HO, Menna-Barreto L. Afternoon School Start Times Are Associated with a Lack of Both Social Jetlag and Sleep Deprivation in Adolescents. J Biol Rhythms. 2020 Aug;35(4):377-390. doi: 10.1177/0748730420927603. Epub 2020 Jun 8. PMID 32508224
- [Background] Crowley SJ, Acebo C, Carskadon MA. Sleep, circadian rhythms, and delayed phase in adolescence. Sleep Med. 2007 Sep;8(6):602-12. doi: 10.1016/j.sleep.2006.12.002. Epub 2007 Mar 26. PMID 17383934
- [Background] Curcio G, Ferrara M, De Gennaro L. Sleep loss, learning capacity and academic performance. Sleep Med Rev. 2006 Oct;10(5):323-37. doi: 10.1016/j.smrv.2005.11.001. Epub 2006 Mar 24. PMID 16564189
- [Background] Dewald JF, Meijer AM, Oort FJ, Kerkhof GA, Bogels SM. The influence of sleep quality, sleep duration and sleepiness on school performance in children and adolescents: A meta-analytic review. Sleep Med Rev. 2010 Jun;14(3):179-89. doi: 10.1016/j.smrv.2009.10.004. Epub 2010 Jan 21. PMID 20093054
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Dijk DJ, Beersma DG, Daan S, Lewy AJ. Bright morning light advances the human circadian system without affecting NREM sleep homeostasis. Am J Physiol. 1989 Jan;256(1 Pt 2):R106-11. doi: 10.1152/ajpregu.1989.256.1.R106. PMID 2912203
- [Background] Durmer JS, Dinges DF. Neurocognitive consequences of sleep deprivation. Semin Neurol. 2005 Mar;25(1):117-29. doi: 10.1055/s-2005-867080. PMID 15798944
- [Background] Dworak M, Schierl T, Bruns T, Struder HK. Impact of singular excessive computer game and television exposure on sleep patterns and memory performance of school-aged children. Pediatrics. 2007 Nov;120(5):978-85. doi: 10.1542/peds.2007-0476. PMID 17974734
- [Background] Fisher PM, Madsen MK, Mc Mahon B, Holst KK, Andersen SB, Laursen HR, Hasholt LF, Siebner HR, Knudsen GM. Three-week bright-light intervention has dose-related effects on threat-related corticolimbic reactivity and functional coupling. Biol Psychiatry. 2014 Aug 15;76(4):332-9. doi: 10.1016/j.biopsych.2013.11.031. Epub 2013 Dec 19. PMID 24439303
- [Background] Gais S, Hullemann P, Hallschmid M, Born J. Sleep-dependent surges in growth hormone do not contribute to sleep-dependent memory consolidation. Psychoneuroendocrinology. 2006 Jul;31(6):786-91. doi: 10.1016/j.psyneuen.2006.02.009. Epub 2006 Apr 18. PMID 16621327
- [Background] Gibson ES, Powles AC, Thabane L, O'Brien S, Molnar DS, Trajanovic N, Ogilvie R, Shapiro C, Yan M, Chilcott-Tanser L. "Sleepiness" is serious in adolescence: two surveys of 3235 Canadian students. BMC Public Health. 2006 May 2;6:116. doi: 10.1186/1471-2458-6-116. PMID 16670019
- [Background] Goel N, Rao H, Durmer JS, Dinges DF. Neurocognitive consequences of sleep deprivation. Semin Neurol. 2009 Sep;29(4):320-39. doi: 10.1055/s-0029-1237117. Epub 2009 Sep 9. PMID 19742409
- [Background] Hatori M, Panda S. The emerging roles of melanopsin in behavioral adaptation to light. Trends Mol Med. 2010 Oct;16(10):435-46. doi: 10.1016/j.molmed.2010.07.005. Epub 2010 Aug 31. PMID 20810319
- [Background] Hysing M, Harvey AG, Linton SJ, Askeland KG, Sivertsen B. Sleep and academic performance in later adolescence: results from a large population-based study. J Sleep Res. 2016 Jun;25(3):318-24. doi: 10.1111/jsr.12373. Epub 2016 Jan 30. PMID 26825591
- [Background] Kopasz M, Loessl B, Hornyak M, Riemann D, Nissen C, Piosczyk H, Voderholzer U. Sleep and memory in healthy children and adolescents - a critical review. Sleep Med Rev. 2010 Jun;14(3):167-77. doi: 10.1016/j.smrv.2009.10.006. Epub 2010 Jan 25. PMID 20093053
- [Background] Kramer Fiala Machado A, Wendt A, Baptista Menezes AM, Goncalves H, Wehrmeister FC. Sleep duration trajectories from adolescence to emerging adulthood: Findings from a population-based birth cohort. J Sleep Res. 2021 Jun;30(3):e13155. doi: 10.1111/jsr.13155. Epub 2020 Aug 17. PMID 32808393
- [Background] Kuula L, Pesonen AK, Merikanto I, Gradisar M, Lahti J, Heinonen K, Kajantie E, Raikkonen K. Development of Late Circadian Preference: Sleep Timing From Childhood to Late Adolescence. J Pediatr. 2018 Mar;194:182-189.e1. doi: 10.1016/j.jpeds.2017.10.068. Epub 2017 Dec 6. PMID 29221693
- [Background] O'Brien LM. The neurocognitive effects of sleep disruption in children and adolescents. Child Adolesc Psychiatr Clin N Am. 2009 Oct;18(4):813-23. doi: 10.1016/j.chc.2009.04.008. PMID 19836689
- [Background] Ortega FB, Ruiz JR, Castillo R, Chillon P, Labayen I, Martinez-Gomez D, Redondo C, Marcos A, Moreno LA; AVENA study group. Sleep duration and cognitive performance in adolescence. The AVENA study. Acta Paediatr. 2010 Mar;99(3):454-6. doi: 10.1111/j.1651-2227.2009.01618.x. Epub 2009 Nov 26. No abstract available. PMID 19958297
- [Background] Pilcher JJ, Walters AS. How sleep deprivation affects psychological variables related to college students' cognitive performance. J Am Coll Health. 1997 Nov;46(3):121-6. doi: 10.1080/07448489709595597. PMID 9394089
- [Background] Randazzo AC, Muehlbach MJ, Schweitzer PK, Walsh JK. Cognitive function following acute sleep restriction in children ages 10-14. Sleep. 1998 Dec 15;21(8):861-8. PMID 9871948
- [Background] Roberts RE, Roberts CR, Duong HT. Sleepless in adolescence: prospective data on sleep deprivation, health and functioning. J Adolesc. 2009 Oct;32(5):1045-57. doi: 10.1016/j.adolescence.2009.03.007. Epub 2009 Apr 9. PMID 19361854
- [Background] Rosenthal NE, Joseph-Vanderpool JR, Levendosky AA, Johnston SH, Allen R, Kelly KA, Souetre E, Schultz PM, Starz KE. Phase-shifting effects of bright morning light as treatment for delayed sleep phase syndrome. Sleep. 1990 Aug;13(4):354-61. PMID 2267478
- [Background] Sadeh A, Gruber R, Raviv A. Sleep, neurobehavioral functioning, and behavior problems in school-age children. Child Dev. 2002 Mar-Apr;73(2):405-17. doi: 10.1111/1467-8624.00414. PMID 11949899
- [Background] Sadeh A, Gruber R, Raviv A. The effects of sleep restriction and extension on school-age children: what a difference an hour makes. Child Dev. 2003 Mar-Apr;74(2):444-55. doi: 10.1111/1467-8624.7402008. PMID 12705565
- [Background] Sadeh A, Raviv A, Gruber R. Sleep patterns and sleep disruptions in school-age children. Dev Psychol. 2000 May;36(3):291-301. doi: 10.1037//0012-1649.36.3.291. PMID 10830974
- [Background] Suratt PM, Barth JT, Diamond R, D'Andrea L, Nikova M, Perriello VA Jr, Carskadon MA, Rembold C. Reduced time in bed and obstructive sleep-disordered breathing in children are associated with cognitive impairment. Pediatrics. 2007 Feb;119(2):320-9. doi: 10.1542/peds.2006-1969. PMID 17272622
- [Background] Walker MP. Cognitive consequences of sleep and sleep loss. Sleep Med. 2008 Sep;9 Suppl 1:S29-34. doi: 10.1016/S1389-9457(08)70014-5. PMID 18929316
- [Background] Wheaton AG, Olsen EO, Miller GF, Croft JB. Sleep Duration and Injury-Related Risk Behaviors Among High School Students--United States, 2007-2013. MMWR Morb Mortal Wkly Rep. 2016 Apr 8;65(13):337-41. doi: 10.15585/mmwr.mm6513a1. PMID 27054407
- [Derived] Teicher MH, Bolger E, Garcia LCH, Hafezi P, Weiser LP, McGreenery CE, Khan A, Ohashi K. Bright light therapy and early morning attention, mathematical performance, electroencephalography and brain connectivity in adolescents with morning sleepiness. PLoS One. 2023 Aug 22;18(8):e0273269. doi: 10.1371/journal.pone.0273269. eCollection 2023. PMID 37607203